CLINICAL TRIAL: NCT05852990
Title: Effect of Glutamine Plus Lactobacillus Reuteri Added to an Astringent Diet in Preventing Diarrhea Caused by Tyrosine Kinase Inhibitors (TKIs) in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Glutamine Plus L. Reuteri Prevents TKI Therapy-diarrhea in Patients With NSCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Head of the Thoracic Oncology Unit and Personalized Medicine Laboratory, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEI/1565/21 INCAN/CEI/0074/22
Record Dates: First submitted 2023-02-24; First posted 2023-05-10 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer With EGFR Mutation
Keywords: Non-Small Cell Lung Cancer; EGFR mutation; Glutamine; Lactobacillus reuteri; standard-care diet
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Glutamine

STUDY DESIGN:
Intervention Model Description: Patients with Non-Small Cell Lung Cancer and EGFR Mutation receiving first or second generation-TKI therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention diet (Experimental): Astringent diet supplemented with one sachet containing 10 grams of glutamine plus 100 million Colony Forming Units (CFU) of Lactobacillus reueri every 12 hours, from baseline treatment up to 6 weeks or death.
  Interventions: Combination Product: Glutamine plus L. reuteri
- Standard diet (No Intervention): Astringent diet from baseline treatment up to 6 weeks or death.

INTERVENTIONS:
Combination Product: Glutamine plus L. reuteri — Glutamine plus Lactobacillus reueri twice daily for up to 6 weeks or death
  Other Names: Glutapak-R
  Arms: Intervention diet

SUMMARY:
This open-label randomized clinical trial aims to evaluate the glutamine plus Lactobacillus reuteri supplementation effect in a standard-of-care diet in EGFR mutant patients with advanced non-small cell lung cancer (NSCLC) under tyrosine kinase inhibitors (TKIs) therapy.

The main question it aims to answer is ¿What is the effect of glutamine plus L. reuteri added to an astringent diet in preventing diarrhea generated by TKI therapy?

Patients will receive an astringent diet supplemented with 10 grams of glutamine and L. reuteri (100 million CFU). Researchers will compare the Glutamine plus L. reuteri diet with a standard astringent diet to see if TKI therapy diarrhea is prevented.

DETAILED DESCRIPTION:
Patients in the experimental group will receive two sachets of Glutapak-R every twelve hours for up to six weeks alongside treating physician-chosen EGFR therapy. Patients in the control group will receive a standard-of-care diet.

All patients will receive nutritional counseling every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* ≥ 18 years old
* Pathologically confirmed diagnosis of NSCLC
* Stage IIIB - IV by the American Joint Committee of Cancer Version 8.
* Candidates to receive EGFR-TKI treatment (1st & 2nd generation TKI)
* ECOG score ≤ 2
* Life expectancy > eight weeks
* Signed written informed consent

Exclusion Criteria:

* Patients who cannot attend the first protocol appointment.
* Treatment with other anti-cancer therapy
* Participating in other clinical trials in the former four weeks
* Any other serious condition or uncontrolled active infection, altered mental status or psychiatric disorder that, in the investigator´s opinion, would limit the ability of an individual to meet the requirements of the study or which affects the interpretability of the results.
* Active hepatitis virus infection (any serotype) or chronic infection with a potential risk of reactivation evaluated through a serological panel.
* Active HIV infection.
* Breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Diarrhea toxicity | every two weeks, from first dose of TKI therapy up to six weeks.
  The diarrhea grade will be determined from 1 to 5 following the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. As shown below:
  grade 1: Increase of < 4 stools per day over baseline; mild increase in ostomy output compared to baseline grade 2: Increase of 4 - 6 stools per day over baseline; moderate increase in ostomy output compared to baseline; limiting instrumental ADL.
  grade 3: Increase of >= 7 stools per day over baseline; hospitalization indicated; severe increase in ostomy output compared to baseline; limiting self-care ADL.
  grade 4: Life-threatening consequences; urgent intervention indicated grade 5: Death
Functional Assessment of Chronic Illness Therapy | Every two weeks, from first dose of TKI therapy up to six weeks.
  This assessment will be evaluated with a specific scale for diarrhea (FACIT instrument), which consists of 11 items that assign a value of 0 to 4 for each one. Higher the score, the better quality of life related to diarrhea.

SECONDARY OUTCOMES:
Grade of gastrointestinal toxicity | Every two weeks, from first dose of TKI therapy up to six weeks.
  This outcome will be determined from grades 1 to 5 according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for gastrointestinal disorders.
Measurement of health related quality of life (QoL) | Every two weeks, from first dose of TKI therapy up to six weeks.
  The QoL of patients with cancer will be determined by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire version 3.0 (EORTC QLQ-C30 v3.0) instrument.
Measurement of quality of life (QoL) for lung cancer patients | Every two weeks, from first dose of TKI therapy up to six weeks.
  The QoL for Lung Cancer patients will be determined by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire version 3.0 (EORTC QLQ-LC13) instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar G Arrieta Rodriguez, M.D., M.Sc., Principal Investigator — Instituto Nacional de Cancerología de México
Locations (1):
- Instituto Nacional de Cancerologia de Mexico, Mexico City, Mexico

REFERENCES:
- [Background] Arrieta O, Nunez-Valencia C, Reynoso-Erazo L, Alvarado S, Flores-Estrada D, Angulo LP, Onate-Ocana LF. Health-related quality of life in patients with lung cancer: validation of the Mexican-Spanish version and association with prognosis of the EORTC QLQ-LC13 questionnaire. Lung Cancer. 2012 Jul;77(1):205-11. doi: 10.1016/j.lungcan.2012.02.005. Epub 2012 Mar 3. PMID 22387006
- [Background] Goldstraw P, Ball D, Jett JR, Le Chevalier T, Lim E, Nicholson AG, Shepherd FA. Non-small-cell lung cancer. Lancet. 2011 Nov 12;378(9804):1727-40. doi: 10.1016/S0140-6736(10)62101-0. Epub 2011 May 10. PMID 21565398
- [Background] Walters S, Maringe C, Coleman MP, Peake MD, Butler J, Young N, Bergstrom S, Hanna L, Jakobsen E, Kolbeck K, Sundstrom S, Engholm G, Gavin A, Gjerstorff ML, Hatcher J, Johannesen TB, Linklater KM, McGahan CE, Steward J, Tracey E, Turner D, Richards MA, Rachet B; ICBP Module 1 Working Group. Lung cancer survival and stage at diagnosis in Australia, Canada, Denmark, Norway, Sweden and the UK: a population-based study, 2004-2007. Thorax. 2013 Jun;68(6):551-64. doi: 10.1136/thoraxjnl-2012-202297. Epub 2013 Feb 11. PMID 23399908
- [Background] Secombe KR, Van Sebille YZA, Mayo BJ, Coller JK, Gibson RJ, Bowen JM. Diarrhea Induced by Small Molecule Tyrosine Kinase Inhibitors Compared With Chemotherapy: Potential Role of the Microbiome. Integr Cancer Ther. 2020 Jan-Dec;19:1534735420928493. doi: 10.1177/1534735420928493. PMID 32493068
- [Background] Achamrah N, Dechelotte P, Coeffier M. Glutamine and the regulation of intestinal permeability: from bench to bedside. Curr Opin Clin Nutr Metab Care. 2017 Jan;20(1):86-91. doi: 10.1097/MCO.0000000000000339. PMID 27749689
- [Background] Sanchez-Lara K, Turcott JG, Juarez E, Guevara P, Nunez-Valencia C, Onate-Ocana LF, Flores D, Arrieta O. Association of nutrition parameters including bioelectrical impedance and systemic inflammatory response with quality of life and prognosis in patients with advanced non-small-cell lung cancer: a prospective study. Nutr Cancer. 2012;64(4):526-34. doi: 10.1080/01635581.2012.668744. Epub 2012 Apr 10. PMID 22489794
- [Background] Arrieta O, Michel Ortega RM, Villanueva-Rodriguez G, Serna-Thome MG, Flores-Estrada D, Diaz-Romero C, Rodriguez CM, Martinez L, Sanchez-Lara K. Association of nutritional status and serum albumin levels with development of toxicity in patients with advanced non-small cell lung cancer treated with paclitaxel-cisplatin chemotherapy: a prospective study. BMC Cancer. 2010 Feb 21;10:50. doi: 10.1186/1471-2407-10-50. PMID 20170547